CLINICAL TRIAL: NCT00223990
Title: A Dbl-blind,Randomized,Controlled,Phase IIb Field Trial in 12-47 Month-old Children in Western Kenya to Eval the Efficacy,Safety and Immunogenicity of the FMP1/AS02A Malaria Vaccine vs Rabies Vaccine
Brief Title: Double-blind, Randomized, Controlled Study of Safety, Immunogenicity and Efficacy of a Candidate Malaria Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); GlaxoSmithKline (Industry); Kenya Medical Research Institute (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: A-13228; IND 9202 (Other: FDA); 1123 (Other: WRAIR)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2020-05-21 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Malaria, Falciparum
Keywords: Plasmodium; falciparum; malaria; vaccine; AS02A adjuvant; FMP1; Merozoite surface protein-1
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Intervention Model Description: Subjects were screened no more than 45 days prior to the first inoculation and were randomized on the first day of vaccination 1:1 between two arms (FMP1/AS02A and rabies vaccine (RabAvert)).
Who Masked: Participant, Investigator
Masking Description: Both study participants and those investigators responsible for evaluation of the endpoints will be blinded as to who receives the test article versus the comparator. On vaccination days, the comparator vaccine will be in the same package as received from the manufacturer. After agitation it will appear clear and pink. The FMP1 antigen and the AS02A adjuvant will be packaged separately. The reconstituted FMPI antigen in the AS02A adjuvant/diluent will have a milky white appearance. Because the vaccines will have a markedly different appearance, contents of the syringe will be concealed as described later in this section. The two vaccine preparation teams, consisting of the study pharmacist, pharmacy assistants, and drug manager (an experienced nurse, clinician, or pharmacist), will be responsible for vaccine preparation. They will also verify that the proper vaccine and vaccine dose is prepared and delivered to each subject.

ARMS (2):
- FMP1/AS02A (Experimental): FMP1/AS02A candidate malaria vaccine was administered IM in the left anterolateral thigh muscle at 0, 1, and 2 months
  Interventions: Biological: FMP1/AS02A
- RabAvert (rabies vaccine) (Active Comparator): RabAvert vaccine was administered IM in the left anterolateral thigh muscle at 0, 1, and 2 months
  Interventions: Biological: RabAvert

INTERVENTIONS:
Biological: FMP1/AS02A — FMP1/AS02A candidate malaria vaccine
  Arms: FMP1/AS02A
Biological: RabAvert — RabAvert rabies vaccine
  Arms: RabAvert (rabies vaccine)

SUMMARY:
This trial is currently evaluating one candidate malaria vaccine, FMP1/AS02A. This candidate malaria vaccine is being developed for the routine immunization of infants and children living in malaria-endemic areas. This vaccine would offer protection against malaria disease due to the parasite Plasmodium falciparum.

Prior to the start of this study, FMP1/AS02A had been given to approximately 60 malaria-naïve adults and 40 adults and 90 children living in malaria-endemic regions.

This study will investigate whether the candidate vaccine prevents malaria disease for 6 months post-vaccination.

One half of the enrolled subjects will receive FMP1/AS02A and the other half rabies vaccine (RabAvert).

DETAILED DESCRIPTION:
Field trial of a candidate antigen/adjuvant conducted at one study center with 12 outlying (satellite) field stations. Subjects were screened no more than 45 days prior to the first inoculation and were randomized on the first day of vaccination 1:1 between two arms (FMP1/AS02A and rabies vaccine). The planned immunization schedule was 0, 1, and 2 months for both study arms; however, the 4-week intervals between doses could be extended for up to 2 additional weeks if temporary suspension was deemed advisable due to serious adverse events (SAEs) or other concerns. Vaccinations were administered intramuscularly (IM) in the left anterolateral thigh muscle unless a compelling reason for using an alternate injection site was evident. Each subject participated in the study approximately 14 months with 7-day follow-up for solicited adverse events (five visits: vaccination day plus post-vaccination days 1, 2, 3, and 6) and 30-day follow-up for unsolicited events (vaccination day plus 29 subsequent days). Follow-up of SAEs continued for study duration. Active case detection occurred during the Efficacy Follow-up Period (169 days, starting 14 days after the third vaccination (Day 71)), active case detection commenced with visits approximately every 28 days to the Walter Reed Project Kombewa clinic and terminated after 6 months (approximately Day 240). The primary study analysis for all endpoints was completed on the cleaned Efficacy Follow-up Period database after a data-lock-point. The Addendum Efficacy Follow-up Period (125 days) started with the end of the Efficacy Follow-up Period (approximately Day 240) and active case detection commenced with visits approximately every 28 days to the Walter Reed Project Kombewa Clinic and terminated after 10 months (approximately Day 364). The study addendum analysis for all endpoints was completed after the Addendum Efficacy Follow-up Period database after a data-lock-point.

Malaria cases were detected actively and passively. Active case detection was handled through scheduled (1) facilitated participant visits to the Kombewa Clinic and (2) field worker visits to participant homes. Passive case detection was handled through unscheduled, self-presentation of participants to the Kombewa Clinic. At scheduled clinic visits, blood samples were taken from all subjects to determine parasite density and hemoglobin levels. At home visits, subjects with fever or other illness within the 24 hours were transported to the clinic for collection of blood samples.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* A healthy male or female child, 12 to 47 months of age on the day of screening
* Written informed consent obtained from at least one parent/guardian before study start
* Available to participate for the study duration (about 14 months)

Exclusion Criteria:

* Acute disease at the time of entry into the study that in the opinion of the investigator may pose a threat to the subject
* Prior receipt of a rabies vaccine or any investigational vaccine
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination. (For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed)
* Administration or anticipated administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid
* Previous vaccination with a vaccine containing MPL or QS21 (e.g., RTS,S/AS02A)
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection. (No HIV test will be performed as part of this study.)
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine components, such as eggs
* History of surgical splenectomy
* Administration of immunoglobulins, blood transfusions, or any other blood products within the six months preceding the first dose of study vaccine or planned administration during the study period
* Simultaneous participation in any other clinical trial
* Acute or chronic cardiovascular, pulmonary, hepatic, or renal condition that in the opinion of the PI, may increase the risk to the subject from participating in the study
* Any other condition or circumstance that in the opinion of the investigator may pose a threat to the subject

Ages: 12 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2005-04-08 (Actual); Primary Completion 2006-04-26 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhards Ogutu, M.D., Principal Investigator — Kenya Medical Research Institute
Locations (1):
- Walter Reed Project, Kombewa Clinic, Kisumu, Nyanza Province, Kenya

REFERENCES:
- [Background] Pichyangkul S, Gettayacamin M, Miller RS, Lyon JA, Angov E, Tongtawe P, Ruble DL, Heppner DG Jr, Kester KE, Ballou WR, Diggs CL, Voss G, Cohen JD, Walsh DS. Pre-clinical evaluation of the malaria vaccine candidate P. falciparum MSP1(42) formulated with novel adjuvants or with alum. Vaccine. 2004 Sep 28;22(29-30):3831-40. doi: 10.1016/j.vaccine.2004.07.023. PMID 15364429
- [Background] Angov E, Aufiero BM, Turgeon AM, Van Handenhove M, Ockenhouse CF, Kester KE, Walsh DS, McBride JS, Dubois MC, Cohen J, Haynes JD, Eckels KH, Heppner DG, Ballou WR, Diggs CL, Lyon JA. Development and pre-clinical analysis of a Plasmodium falciparum Merozoite Surface Protein-1(42) malaria vaccine. Mol Biochem Parasitol. 2003 May;128(2):195-204. doi: 10.1016/s0166-6851(03)00077-x. PMID 12742586
- [Derived] Ogutu BR, Apollo OJ, McKinney D, Okoth W, Siangla J, Dubovsky F, Tucker K, Waitumbi JN, Diggs C, Wittes J, Malkin E, Leach A, Soisson LA, Milman JB, Otieno L, Holland CA, Polhemus M, Remich SA, Ockenhouse CF, Cohen J, Ballou WR, Martin SK, Angov E, Stewart VA, Lyon JA, Heppner DG, Withers MR; MSP-1 Malaria Vaccine Working Group. Blood stage malaria vaccine eliciting high antigen-specific antibody concentrations confers no protection to young children in Western Kenya. PLoS One. 2009;4(3):e4708. doi: 10.1371/journal.pone.0004708. Epub 2009 Mar 5. PMID 19262754

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened no more than 45 days prior to the first inoculation and were randomized on the first day of vaccination 1:1 between two arms (FMP1/AS02A and rabies vaccine) at the Walter Reed Project Kombewa Clinic in Kombewa Division, Kisumu District, Nyanze Province, Western Kenya (and 12 small field stations within Kombewa Division).
Period: Overall Study
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Started | 200 | 200
Completed | 193 | 191
Not Completed | 7 | 9
Not completed — Moved from area | 2 | 1
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine) | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: Months] — Population: Demographics were reported per field station
  Months
    Walter Reed Project Field Station: number analyzed (Participants) | 43 | 45 | 88
    Walter Reed Project Field Station | 28.6 (10.6) | 29.2 (10.9) | 28.9 (10.7)
    Abol Field Station: number analyzed (Participants) | 14 | 12 | 26
    Abol Field Station | 34.3 (9.7) | 28.9 (10.0) | 31.6 (10.0)
    Bar-Korwa Field Station: number analyzed (Participants) | 7 | 5 | 12
    Bar-Korwa Field Station | 22.0 (6.2) | 32.8 (5.9) | 26.6 (8.0)
    Got-Aglu Field Station: number analyzed (Participants) | 15 | 17 | 32
    Got-Aglu Field Station | 29.1 (11.8) | 25.0 (8.6) | 26.8 (10.2)
    Kitare Field Station: number analyzed (Participants) | 19 | 17 | 36
    Kitare Field Station | 30.2 (10.7) | 29.9 (10.0) | 30.1 (10.2)
    Kuoyo-Kowe Field Station: number analyzed (Participants) | 17 | 18 | 35
    Kuoyo-Kowe Field Station | 31.1 (9.3) | 31.7 (9.4) | 31.4 (9.2)
    Manyanda Field Station: number analyzed (Participants) | 8 | 8 | 16
    Manyanda Field Station | 30.6 (6.4) | 31.1 (8.2) | 30.9 (7.0)
    Mirieri Field Station: number analyzed (Participants) | 18 | 12 | 30
    Mirieri Field Station | 30.3 (10.0) | 26.5 (10.1) | 28.8 (10.0)
    Nduru Field Station: number analyzed (Participants) | 10 | 15 | 25
    Nduru Field Station | 26.1 (10.2) | 34.6 (10.2) | 30.9 (10.9)
    Oruga Field Station: number analyzed (Participants) | 19 | 20 | 39
    Oruga Field Station | 30.5 (9.5) | 33.1 (9.6) | 31.8 (9.5)
    Osewre Field Station: number analyzed (Participants) | 12 | 9 | 21
    Osewre Field Station | 31.1 (11.3) | 30.7 (8.4) | 30.9 (9.8)
    Ranen Field Station: number analyzed (Participants) | 11 | 12 | 23
    Ranen Field Station | 26.2 (10.9) | 32.2 (11.2) | 29.5 (11.2)
    Reru Field Station: number analyzed (Participants) | 7 | 10 | 17
    Reru Field Station | 26.9 (11.0) | 30.3 (10.8) | 28.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographics were reported per field station.
  193 participants completed the study in the FMP1/AS02A arm.
  191 participants completed the study in the RabAvert arm.
  Participants
    WRAIR Field Station: number analyzed (Participants) | 41 | 41 | 82
    WRAIR Field Station: Female | 16 | 17 | 33
    WRAIR Field Station: Male | 25 | 24 | 49
    Abol Field Station: number analyzed (Participants) | 14 | 12 | 26
    Abol Field Station: Female | 7 | 4 | 11
    Abol Field Station: Male | 7 | 8 | 15
    Bar-Korwa Field Station: number analyzed (Participants) | 7 | 5 | 12
    Bar-Korwa Field Station: Female | 3 | 3 | 6
    Bar-Korwa Field Station: Male | 4 | 2 | 6
    Got-Aglu Field Station: number analyzed (Participants) | 14 | 17 | 31
    Got-Aglu Field Station: Female | 6 | 6 | 12
    Got-Aglu Field Station: Male | 8 | 11 | 19
    Kitare Field Station: number analyzed (Participants) | 19 | 17 | 36
    Kitare Field Station: Female | 10 | 5 | 15
    Kitare Field Station: Male | 9 | 12 | 21
    Kuoyo-Kowe Field Station: number analyzed (Participants) | 17 | 18 | 35
    Kuoyo-Kowe Field Station: Female | 8 | 7 | 15
    Kuoyo-Kowe Field Station: Male | 9 | 11 | 20
    Manyanda Field Station: number analyzed (Participants) | 8 | 7 | 15
    Manyanda Field Station: Female | 5 | 5 | 10
    Manyanda Field Station: Male | 3 | 2 | 5
    Mirieri Field Station: number analyzed (Participants) | 18 | 11 | 29
    Mirieri Field Station: Female | 13 | 3 | 16
    Mirieri Field Station: Male | 5 | 8 | 13
    Nduru Kadero Field Station: number analyzed (Participants) | 10 | 13 | 23
    Nduru Kadero Field Station: Female | 8 | 5 | 13
    Nduru Kadero Field Station: Male | 2 | 8 | 10
    Oruga Field Station: number analyzed (Participants) | 19 | 18 | 37
    Oruga Field Station: Female | 7 | 7 | 14
    Oruga Field Station: Male | 12 | 11 | 23
    Osewre Field Station: number analyzed (Participants) | 11 | 9 | 20
    Osewre Field Station: Female | 3 | 6 | 9
    Osewre Field Station: Male | 8 | 3 | 11
    Ranen Field Station: number analyzed (Participants) | 10 | 12 | 22
    Ranen Field Station: Female | 6 | 5 | 11
    Ranen Field Station: Male | 4 | 7 | 11
    Reru Field Station: number analyzed (Participants) | 7 | 10 | 17
    Reru Field Station: Female | 5 | 5 | 10
    Reru Field Station: Male | 2 | 5 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Kenya | 200 | 200 | 400
Malaria Prevention - WRAIR Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the WRAIR Field Station Population: Study specific baseline measures were presented per field station. 82 patients were randomized at this field station.
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 41 | 41 | 82
    Always sleep under mosquito net | 34 | 31 | 65
    Use topical mosquito repellents: number analyzed (Participants) | 41 | 41 | 82
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 41 | 41 | 82
    Use mosquito coils or sprays | 6 | 7 | 13
    Other: number analyzed (Participants) | 41 | 41 | 82
    Other | 0 | 0 | 0
Hemoglobin, g/dL - WRAIR Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values for subjects at the WRAIR Field Station Population: Study specific baseline measures were presented per field station. 82 patients were randomized at this field station.
  g/dL
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 1.16 (1.377) | 10.53 (1.18) | 10.40 (1.29)
Sickle Cell Status - WRAIR Field Station [Count of Participants; unit: Participants] — Participants at the WRAIR Field Station were analyzed for Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 82 participants were randomized at this field station. However, only 73 participants were analyzed for Sickle Cell Status and G6PD Deficiency.
  Participants
    AA: number analyzed (Participants) | 41 | 41 | 82
    AA | 37 | 36 | 73
    AS: number analyzed (Participants) | 41 | 41 | 82
    AS | 3 | 5 | 8
    AD: number analyzed (Participants) | 41 | 41 | 82
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 41 | 41 | 82
    A+ Hb Kenya | 1 | 0 | 1
    G6PD deficient: number analyzed (Participants) | 41 | 41 | 82
    G6PD deficient | 4 | 6 | 10
Alpha-Thalassemia - WRAIR Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the WRAIR Field Station Population: Study specific baseline measures were presented per field station. 82 patients were randomized at this field station.
  Participants
    Hetero: number analyzed (Participants) | 41 | 41 | 82
    Hetero | 17 | 20 | 37
    Normal: number analyzed (Participants) | 41 | 41 | 82
    Normal | 21 | 20 | 41
    Homo: number analyzed (Participants) | 41 | 41 | 82
    Homo | 3 | 1 | 4
Parasite Density (par/µL blood) - WRAIR Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the WRAIR Field Station Population: Study specific baseline measures were presented per field station. 82 patients were randomized at this field station.
  par/µL blood
    number analyzed (Participants) | 41 | 41 | 82
    (all) | 5045.3 (13280.0) | 5716.3 (24832.9) | 5380.8 (19792.3)
Malaria Prevention - Abol Field Station [Count of Participants; unit: Participants] — Baseline Malaria prevention practiced by subjects at the Abol Field Station Population: Study specific baseline measures were presented per field station. 26 patients were randomized at this field station.
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 14 | 12 | 26
    Always sleep under mosquito net | 11 | 11 | 22
    Use topical mosquito repellents: number analyzed (Participants) | 14 | 12 | 26
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 14 | 12 | 26
    Use mosquito coils or sprays | 1 | 1 | 2
    Other: number analyzed (Participants) | 14 | 12 | 26
    Other | 0 | 0 | 0
Hemoglobin, g/dL - Abol Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Abol Field Station Population: Study specific baseline measures were presented per field station. 26 patients were randomized at this field station.
  g/dL
    number analyzed (Participants) | 14 | 12 | 26
    (all) | 10.69 (0.70) | 9.99 (1.13) | 10.37 (0.98)
Sickle Cell Status - Abol Field Station [Count of Participants; unit: Participants] — Participants at the Abol Field Station were analyzed for Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 26 patients were randomized at this field station.
  Participants
    AA: number analyzed (Participants) | 14 | 12 | 26
    AA | 12 | 7 | 19
    AS: number analyzed (Participants) | 14 | 12 | 26
    AS | 2 | 4 | 6
    AD: number analyzed (Participants) | 14 | 12 | 26
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 14 | 12 | 26
    A+ Hb Kenya | 0 | 1 | 1
    G6PD deficient: number analyzed (Participants) | 14 | 12 | 26
    G6PD deficient | 0 | 1 | 1
Baseline Alpha-Thalassemia - Abol Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Abol Field Station Population: Study specific baseline measures were presented per field station. 26 patients were randomized at this field station.
  Participants
    Hetero: number analyzed (Participants) | 14 | 12 | 26
    Hetero | 6 | 3 | 9
    Normal: number analyzed (Participants) | 14 | 12 | 26
    Normal | 7 | 8 | 15
    Homo: number analyzed (Participants) | 14 | 12 | 26
    Homo | 1 | 1 | 2
Baseline Density (par-µL blood)- Abol Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the Abol Field Station Population: Study specific baseline measures were presented per field station. 26 patients were randomized at this field station.
  par/µL blood
    number analyzed (Participants) | 14 | 12 | 26
    (all) | 1509.6 (2816.8) | 303.5 (754.7) | 963.0 (2180.0)
Baseline Malaria Prevention - Bar-Korwa Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Bar-Korwa Field Station Population: Study specific baseline measures were presented per field station. 12 patients were randomized at this field station.
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 7 | 5 | 12
    Always sleep under mosquito net | 7 | 5 | 12
    Use topical mosquito repellents: number analyzed (Participants) | 7 | 5 | 12
    Use topical mosquito repellents | 0 | 0 | 0
    Use moquito coils or sprays: number analyzed (Participants) | 7 | 5 | 12
    Use moquito coils or sprays | 0 | 1 | 1
    Other: number analyzed (Participants) | 7 | 5 | 12
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Bar-Korwa Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values for subjects at the Bar-Korwa Field Station Population: Study specific baseline measures were presented per field station. 12 patients were randomized at this field station.
  g/dL
    number analyzed (Participants) | 7 | 5 | 12
    (all) | 10.24 (0.91) | 10.28 (0.84) | 10.26 (0.84)
Baseline Sickle Cell Status - Bar-Korwa Field Station [Count of Participants; unit: Participants] — Participants at the Bar-Korwa Field Station were analyzed for baseline Sickle Cell status and G6PD Deficiency Population: Study specific baseline measures were presented per field station. 12 patients were randomized at this field station.
  Participants
    AA: number analyzed (Participants) | 7 | 5 | 12
    AA | 3 | 4 | 7
    AS: number analyzed (Participants) | 7 | 5 | 12
    AS | 4 | 1 | 5
    AD: number analyzed (Participants) | 7 | 5 | 12
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 7 | 5 | 12
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 7 | 5 | 12
    G6PD deficient | 0 | 1 | 1
Baseline Alpha-Thalassemia- Bar-Korwa Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Bar-Korwa Field Station Population: Study specific baseline measures were presented per field station. 12 patients were randomized at this field station.
  Participants
    Hetero: number analyzed (Participants) | 7 | 5 | 12
    Hetero | 0 | 2 | 2
    Normal: number analyzed (Participants) | 7 | 5 | 12
    Normal | 6 | 3 | 9
    Homo: number analyzed (Participants) | 7 | 5 | 12
    Homo | 1 | 0 | 1
Baseline Parasite Density (par/µL blood) - Bar-Korwa Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Bar-Korwa Field Station Population: Study specific baseline measures were presented per field station. 12 patients were randomized at this field station.
  par/µL
    number analyzed (Participants) | 7 | 5 | 12
    (all) | 1481.1 (3918.5) | 1679.0 (2907.7) | 1563.5 (3385.3)
Baseline Malaria Prevention - Got-Aglu Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Got-Aglu Field Station Population: Study specific baseline measures were presented per field station. 31patients were randomized at this field station.
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 14 | 17 | 31
    Always sleep under mosquito net | 8 | 8 | 16
    Use topical mosquito repellents: number analyzed (Participants) | 14 | 17 | 31
    Use topical mosquito repellents | 1 | 0 | 1
    Use mosquito coils or sprays: number analyzed (Participants) | 14 | 17 | 31
    Use mosquito coils or sprays | 4 | 7 | 11
    Other: number analyzed (Participants) | 14 | 17 | 31
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Got-Aglu Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Got-Aglu Field Station Population: Study specific baseline measures were presented per field station. 31patients were randomized at this field station.
  g/dL
    number analyzed (Participants) | 14 | 17 | 31
    (all) | 10.42 (1.36) | 10.30 (1.38) | 10.35 (1.35)
Baseline Sickle Cell Status - Got-Aglu Field Station [Count of Participants; unit: Participants] — Participants at the Got-Aglu Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 31patients were randomized at this field station.
  Participants
    AA: number analyzed (Participants) | 14 | 17 | 31
    AA | 8 | 14 | 22
    AS: number analyzed (Participants) | 14 | 17 | 31
    AS | 5 | 3 | 8
    AD: number analyzed (Participants) | 14 | 17 | 31
    AD | 1 | 0 | 1
    A+ Hb Kenya: number analyzed (Participants) | 14 | 17 | 31
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 14 | 17 | 31
    G6PD deficient | 2 | 3 | 5
Baseline Alpha-Thalassemia - Got-Aglu Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Got-Aglu Field Station Population: Study specific baseline measures were presented per field station. 31patients were randomized at this field station.
  Participants
    Hetero: number analyzed (Participants) | 14 | 17 | 31
    Hetero | 9 | 10 | 19
    Normal: number analyzed (Participants) | 14 | 17 | 31
    Normal | 4 | 6 | 10
    Homo: number analyzed (Participants) | 14 | 17 | 31
    Homo | 1 | 1 | 2
Baseline Parasite Density (par/µL blood) - Got-Aglu Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Got-Aglu Field Station Population: Study specific baseline measures were presented per field station. 31patients were randomized at this field station.
  par/µL
    number analyzed (Participants) | 14 | 17 | 31
    (all) | 2427.1 (6899.7) | 3932.5 (7509.3) | 3252.7 (7161.3)
Baseline Malarie Prevention - Kitare Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Kitare Field Station Population: Study specific baseline measures were presented per field station. 36 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 19 | 17 | 36
    Always sleep under mosquito net | 17 | 16 | 33
    Use topical mosquito repellents: number analyzed (Participants) | 19 | 17 | 36
    Use topical mosquito repellents | 1 | 0 | 1
    Use mosquito coils or sprays: number analyzed (Participants) | 19 | 17 | 36
    Use mosquito coils or sprays | 0 | 1 | 1
    Other: number analyzed (Participants) | 19 | 17 | 36
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Kitare Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Kitare Field Station Population: Study specific baseline measures were presented per field station. 36 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 19 | 17 | 36
    (all) | 10.42 (1.10) | 9.96 (0.94) | 10.20 (1.04)
Baseline Sickle Cell Status - Kitare Field Station [Count of Participants; unit: Participants] — Participants at the Kitare Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 36 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 19 | 17 | 36
    AA | 14 | 10 | 24
    AS: number analyzed (Participants) | 19 | 17 | 36
    AS | 5 | 7 | 12
    AD: number analyzed (Participants) | 19 | 17 | 36
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 19 | 17 | 36
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 19 | 17 | 36
    G6PD deficient | 1 | 2 | 3
Baseline Alpha-Thalassemia - Kitare Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Kitare Field Station Population: Study specific baseline measures were presented per field station. 36 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 19 | 17 | 36
    Hetero | 9 | 10 | 19
    Normal: number analyzed (Participants) | 19 | 17 | 36
    Normal | 7 | 6 | 13
    Homo: number analyzed (Participants) | 19 | 17 | 36
    Homo | 3 | 1 | 4
Baseline Parasite Density (par/µL blood) - Kitare Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Kitare Field Station Population: Study specific baseline measures were presented per field station. 36 patients were randomized at this field station
  par/µL
    number analyzed (Participants) | 19 | 17 | 36
    (all) | 1645.5 (4375.6) | 550.1 (1416.7) | 1144.8 (3355.7)
Baseline Malaria Prevention - Kuoyo-Kowe Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Kuoyo-Kowe Field Station Population: Study specific baseline measures were presented per field station. 35 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 17 | 18 | 35
    Always sleep under mosquito net | 9 | 12 | 21
    Use topical mosquito repellents: number analyzed (Participants) | 17 | 18 | 35
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 17 | 18 | 35
    Use mosquito coils or sprays | 3 | 4 | 7
    Other: number analyzed (Participants) | 17 | 18 | 35
    Other | 1 | 0 | 1
Baseline Hemoglobin (g/dL) - Kuoyo-Kowe Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Kuoyo-Kowe Field Station Population: Study specific baseline measures were presented per field station. 35 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 10.75 (1.20) | 10.19 (1.28) | 10.46 (1.25)
Baseline Sickle Cell Status - Kuoyo-Kowe Field Station [Count of Participants; unit: Participants] — Participants at the Kuoyo-Kowe Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 35 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 17 | 18 | 35
    AA | 13 | 16 | 29
    AS: number analyzed (Participants) | 17 | 18 | 35
    AS | 4 | 2 | 6
    AD: number analyzed (Participants) | 17 | 18 | 35
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 17 | 18 | 35
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 17 | 18 | 35
    G6PD deficient | 5 | 2 | 7
Baseline Alpha-Thalassemia - Kuoyo-Kowe Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Kuoyo-Kowe Field Station Population: Study specific baseline measures were presented per field station. 35 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 17 | 18 | 35
    Hetero | 3 | 8 | 11
    Normal: number analyzed (Participants) | 17 | 18 | 35
    Normal | 13 | 7 | 20
    Homo: number analyzed (Participants) | 17 | 18 | 35
    Homo | 1 | 3 | 4
Baseline Parasite Density (par/µL blood) - Kuoyo-Kowe Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Kuoyo-Kowe Field Station Population: Study specific baseline measures were presented per field station. 35 patients were randomized at this field station
  par/µL
    number analyzed (Participants) | 17 | 18 | 35
    (all) | 1073.0 (2664.) | 1185.0 (4230.4) | 1130.6 (3502.5)
Baseline Malaria Prevention - Manyanda Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Manyanda Field Station Population: Study specific baseline measures were presented per field station. 15 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 8 | 7 | 15
    Always sleep under mosquito net | 7 | 6 | 13
    Use topical mosquito repellents: number analyzed (Participants) | 8 | 7 | 15
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 8 | 7 | 15
    Use mosquito coils or sprays | 2 | 1 | 3
    Other: number analyzed (Participants) | 8 | 7 | 15
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Manyanda Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Manyanda Field Station Population: Study specific baseline measures were presented per field station. 15 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 8 | 7 | 15
    (all) | 10.34 (1.29) | 10.46 (7.67) | 10.39 (1.42)
Baseline Sick Cell Status - Manyanda Field Station [Count of Participants; unit: Participants] — Participants at the Manyanda Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 15 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 8 | 7 | 15
    AA | 6 | 4 | 10
    AS: number analyzed (Participants) | 8 | 7 | 15
    AS | 2 | 3 | 5
    AD: number analyzed (Participants) | 8 | 7 | 15
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 8 | 7 | 15
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 8 | 7 | 15
    G6PD deficient | 0 | 0 | 0
Baseline Alpha-Thalassemia - Manyanda Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Manyanda Field Station Population: Study specific baseline measures were presented per field station. 15 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 8 | 7 | 15
    Hetero | 3 | 1 | 4
    Normal: number analyzed (Participants) | 8 | 7 | 15
    Normal | 5 | 6 | 11
    Homo: number analyzed (Participants) | 8 | 7 | 15
    Homo | 0 | 0 | 0
Baseline Parasite Density (par/µL blood) - Manyanda Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Manyanda Field Station Population: Study specific baseline measures were presented per field station. 15 patients were randomized at this field station
  par/µL
    number analyzed (Participants) | 8 | 7 | 15
    (all) | 148.9 (330.1) | 2441.0 (4236.4) | 1218.5 (3024.4)
Baseline Malaria Prevention - Mirieri Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Mirieri Field Station Population: Study specific baseline measures were presented per field station. 29 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 18 | 11 | 29
    Always sleep under mosquito net | 10 | 6 | 16
    Use topical mosquito repellents: number analyzed (Participants) | 18 | 11 | 29
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 18 | 11 | 29
    Use mosquito coils or sprays | 1 | 3 | 4
    Other: number analyzed (Participants) | 18 | 11 | 29
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Mirieri Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Mirieri Field Station Population: Study specific baseline measures were presented per field station. 29 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 18 | 11 | 29
    (all) | 11.10 (0.97) | 10.48 (1.38) | 10.87 (1.16)
Baseline Sickle Cell Status - Mirieri Field Station [Count of Participants; unit: Participants] — Participants at the Mirieri Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 29 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 18 | 11 | 29
    AA | 16 | 8 | 24
    AS: number analyzed (Participants) | 18 | 11 | 29
    AS | 2 | 3 | 5
    AD: number analyzed (Participants) | 18 | 11 | 29
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 18 | 11 | 29
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 18 | 11 | 29
    G6PD deficient | 3 | 0 | 3
Baseline Alpha-Thalassemia - Mirieri Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Mirieri Field Station Population: Study specific baseline measures were presented per field station. 29 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 18 | 11 | 29
    Hetero | 8 | 6 | 14
    Normal: number analyzed (Participants) | 18 | 11 | 29
    Normal | 8 | 4 | 12
    Homo: number analyzed (Participants) | 18 | 11 | 29
    Homo | 2 | 1 | 3
Baseline Parasite Density (par/µL blood) - Mirieri Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Mirieri Field Station Population: Study specific baseline measures were presented per field station. 29 patients were randomized at this field station
  par/µL
    number analyzed (Participants) | 18 | 11 | 29
    (all) | 1669.4 (3848.2) | 15775 (51756.8) | 7019.6 (31662.4)
Baseline Malaria Prevention - Nduru Kadero Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Nduru Kadero Field Station Population: Study specific baseline measures were presented per field station. 23 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 10 | 13 | 23
    Always sleep under mosquito net | 5 | 8 | 13
    Use topical mosquito repellents: number analyzed (Participants) | 10 | 13 | 23
    Use topical mosquito repellents | 1 | 0 | 1
    Use mosquito coils or sprays: number analyzed (Participants) | 10 | 13 | 23
    Use mosquito coils or sprays | 5 | 2 | 7
    Other: number analyzed (Participants) | 10 | 13 | 23
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Nduru Kadero Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Nduru Kadero Field Station Population: Study specific baseline measures were presented per field station. 23 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 10 | 13 | 23
    (all) | 10.48 (1.18) | 10.78 (1.28) | 10.66 (1.21)
Baseline Sickle Cell Status - Nduru Kadero Field Station [Count of Participants; unit: Participants] — Participants at the Nduru Kadero Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 23 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 10 | 13 | 23
    AA | 9 | 11 | 20
    AS: number analyzed (Participants) | 10 | 13 | 23
    AS | 1 | 2 | 3
    AD: number analyzed (Participants) | 10 | 13 | 23
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 10 | 13 | 23
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 10 | 13 | 23
    G6PD deficient | 0 | 1 | 1
Baseline Alpha-Thalassemia - Nduru Kadero Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Nduru Kadero Field Station Population: Study specific baseline measures were presented per field station. 23 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 10 | 13 | 23
    Hetero | 5 | 10 | 15
    Normal: number analyzed (Participants) | 10 | 13 | 23
    Normal | 4 | 2 | 6
    Homo: number analyzed (Participants) | 10 | 13 | 23
    Homo | 1 | 1 | 2
Baseline Parasite Density (par/µL blood) - Nduru Kadero Field Station [Mean (Standard Deviation); unit: par/µL] — Baseline Parasite Density values (par/µL blood) for subjects at the Nduru Kadero Field Station Population: Study specific baseline measures were presented per field station. 23 patients were randomized at this field station
  par/µL
    number analyzed (Participants) | 10 | 13 | 23
    (all) | 1676.5 (5123.2) | 6749.7 (20674.1) | 4543.9 (15826.8)
Baseline Malaria Prevention - Oruga Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Oruga Field Station Population: Study specific baseline measures were presented per field station. 37 patients were randomized at this field station
  Participants
    Alwasy sleep under mosquito net: number analyzed (Participants) | 19 | 18 | 37
    Alwasy sleep under mosquito net | 15 | 12 | 27
    Use topical mosquito repellents: number analyzed (Participants) | 19 | 18 | 37
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 19 | 18 | 37
    Use mosquito coils or sprays | 1 | 3 | 4
    Other: number analyzed (Participants) | 19 | 18 | 37
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Oruga Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Oruga Field Station Population: Study specific baseline measures were presented per field station. 37 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 10.57 (1.00) | 9.96 (1.23) | 10.27 (1.15)
Baseline Sickle Cell Status - Oruga Field Station [Count of Participants; unit: Participants] — Participants at the Oruga Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 37 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 19 | 18 | 37
    AA | 15 | 16 | 31
    AS: number analyzed (Participants) | 19 | 18 | 37
    AS | 3 | 2 | 5
    AD: number analyzed (Participants) | 19 | 18 | 37
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 19 | 18 | 37
    A+ Hb Kenya | 1 | 0 | 1
    G6PD deficient: number analyzed (Participants) | 19 | 18 | 37
    G6PD deficient | 2 | 2 | 4
Baseline Alpha-Thalassemia - Oruga Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Oruga Field Station Population: Study specific baseline measures were presented per field station. 37 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 19 | 18 | 37
    Hetero | 4 | 7 | 11
    Normal: number analyzed (Participants) | 19 | 18 | 37
    Normal | 10 | 9 | 19
    Homo: number analyzed (Participants) | 19 | 18 | 37
    Homo | 5 | 2 | 7
Baseline Parasite Density (par/µL blood) - Oruga Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the Oruga Field Station Population: Study specific baseline measures were presented per field station. 37 patients were randomized at this field station
  par/µL blood
    number analyzed (Participants) | 19 | 18 | 37
    (all) | 1481.6 (3068.2) | 3034.9 (5151.7) | 2237.3 (4226.0)
Baseline Malaria Prevention - Osewre Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Osewre Field Station Population: Study specific baseline measures were presented per field station. 20 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 11 | 9 | 20
    Always sleep under mosquito net | 8 | 6 | 14
    Use topical mosquito repellents: number analyzed (Participants) | 11 | 9 | 20
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 11 | 9 | 20
    Use mosquito coils or sprays | 2 | 1 | 3
    Other: number analyzed (Participants) | 11 | 9 | 20
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Osewre Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Osewre Field Station Population: Study specific baseline measures were presented per field station. 20 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 10.06 (1.62) | 10.18 (1.08) | 10.12 (1.37)
Baseline Sickle Cell Status - Osewre Field Station [Count of Participants; unit: Participants] — Participants at the Osewre Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 20 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 11 | 9 | 20
    AA | 11 | 9 | 20
    AS: number analyzed (Participants) | 11 | 9 | 20
    AS | 0 | 0 | 0
    AD: number analyzed (Participants) | 11 | 9 | 20
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 11 | 9 | 20
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 11 | 9 | 20
    G6PD deficient | 0 | 2 | 2
Baseline Alpha-Thalassemia - Osewre Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Osewre Field Station Population: Study specific baseline measures were presented per field station. 20 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 11 | 9 | 20
    Hetero | 3 | 5 | 8
    Normal: number analyzed (Participants) | 11 | 9 | 20
    Normal | 8 | 3 | 11
    Homo: number analyzed (Participants) | 11 | 9 | 20
    Homo | 0 | 1 | 1
Baseline Parasite Density (par/µL blood) - Osewre Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the Osewre Field Station Population: Study specific baseline measures were presented per field station. 20 patients were randomized at this field station
  par/µL blood
    number analyzed (Participants) | 11 | 9 | 20
    (all) | 5288.3 (10961.1) | 1129.7 (2548.3) | 3416.9 (8394.9)
Baseline Malaria Prevention - Ranen Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Ranen Field Station Population: Study specific baseline measures were presented per field station. 22 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 10 | 12 | 22
    Always sleep under mosquito net | 5 | 12 | 17
    Use topical mosquito repellents: number analyzed (Participants) | 10 | 12 | 22
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 10 | 12 | 22
    Use mosquito coils or sprays | 3 | 0 | 3
    Other: number analyzed (Participants) | 10 | 12 | 22
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Ranen Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Ranen Field Station Population: Study specific baseline measures were presented per field station. 22 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 10 | 12 | 22
    (all) | 10.01 (1.03) | 10.34 (1.24) | 10.19 (1.14)
Baseline Sickle Cell Status - Ranen Field Station [Count of Participants; unit: Participants] — Participants at the Ranen Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 22 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 10 | 12 | 22
    AA | 9 | 9 | 18
    AS: number analyzed (Participants) | 10 | 12 | 22
    AS | 1 | 3 | 4
    AD: number analyzed (Participants) | 10 | 12 | 22
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 10 | 12 | 22
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 10 | 12 | 22
    G6PD deficient | 1 | 1 | 2
Baseline Alpha-Thalassemia - Ranen Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Ranen Field Station Population: Study specific baseline measures were presented per field station. 22 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 10 | 12 | 22
    Hetero | 6 | 5 | 11
    Normal: number analyzed (Participants) | 10 | 12 | 22
    Normal | 2 | 6 | 8
    Homo: number analyzed (Participants) | 10 | 12 | 22
    Homo | 2 | 1 | 3
Baseline Parasite Density (par/µL blood) - Ranen Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the Ranen Field Station Population: Study specific baseline measures were presented per field station. 22 patients were randomized at this field station
  par/µL blood
    number analyzed (Participants) | 10 | 12 | 22
    (all) | 3734.0 (11675.1) | 5906.4 (14161.9) | 4871.9 (12761.4)
Baseline Malaria Prevention - Reru Field Station [Count of Participants; unit: Participants] — Baseline malaria prevention practiced by subjects at the Reru Field Station Population: Study specific baseline measures were presented per field station. 17 patients were randomized at this field station
  Participants
    Always sleep under mosquito net: number analyzed (Participants) | 7 | 10 | 17
    Always sleep under mosquito net | 3 | 7 | 10
    Use topical mosquito repellents: number analyzed (Participants) | 7 | 10 | 17
    Use topical mosquito repellents | 0 | 0 | 0
    Use mosquito coils or sprays: number analyzed (Participants) | 7 | 10 | 17
    Use mosquito coils or sprays | 3 | 5 | 8
    Other: number analyzed (Participants) | 7 | 10 | 17
    Other | 0 | 0 | 0
Baseline Hemoglobin (g/dL) - Reru Field Station [Mean (Standard Deviation); unit: g/dL] — Baseline Hemoglobin values (g/dL) for subjects at the Reru Field Station Population: Study specific baseline measures were presented per field station. 17 patients were randomized at this field station
  g/dL
    number analyzed (Participants) | 7 | 10 | 17
    (all) | 10.44 (1.57) | 10.14 (1.03) | 10.26 (1.24)
Baseline Sickle Cell Status - Reru Field Station [Count of Participants; unit: Participants] — Participants at the Reru Field Station were analyzed for baseline Sickle Cell status and G6PD deficiency Population: Study specific baseline measures were presented per field station. 17 patients were randomized at this field station
  Participants
    AA: number analyzed (Participants) | 7 | 10 | 17
    AA | 5 | 8 | 13
    AS: number analyzed (Participants) | 7 | 10 | 17
    AS | 2 | 2 | 4
    AD: number analyzed (Participants) | 7 | 10 | 17
    AD | 0 | 0 | 0
    A+ Hb Kenya: number analyzed (Participants) | 7 | 10 | 17
    A+ Hb Kenya | 0 | 0 | 0
    G6PD deficient: number analyzed (Participants) | 7 | 10 | 17
    G6PD deficient | 2 | 2 | 4
Baseline Alpha-Thalassemia - Reru Field Station [Count of Participants; unit: Participants] — Baseline Alpha-Thalassemia values for subjects at the Reru Field Station Population: Study specific baseline measures were presented per field station. 17 patients were randomized at this field station
  Participants
    Hetero: number analyzed (Participants) | 7 | 10 | 17
    Hetero | 4 | 5 | 9
    Normal: number analyzed (Participants) | 7 | 10 | 17
    Normal | 2 | 4 | 6
    Homo: number analyzed (Participants) | 7 | 10 | 17
    Homo | 1 | 1 | 2
Baseline Parasite Density (par/µL blood) - Reru Field Station [Mean (Standard Deviation); unit: par/µL blood] — Baseline Parasite Density values (par/µL blood) for subjects at the Reru Field Station Population: Study specific baseline measures were presented per field station. 17 patients were randomized at this field station
  par/µL blood
    number analyzed (Participants) | 7 | 10 | 17
    (all) | 823.5 (1490.1) | 5377.5 (13315.9) | 3502.3 (10291.2)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Time to First Clinical Episode of P Falciparum Malaria During the Efficacy Follow-up Period Adjusted for Time at Risk - Intent to Treat (ITT) Population
Description: Days to first clinical episode of P falciparum malaria during the efficacy f/u period for ITT population
  Time at Risk adjusted for:
  SA= study absence MT= malaria treatment SA MT= study absence and malaria treatment
  Case Definitions:
  Primary = >37.5°C with presence of a density of asexual stage P. falciparum >50K parasites/µL blood Secondary (200) = >37.5°C with presence of a density of asexual stage P. falciparum >200K parasites/µL blood Secondary (100) = >37.5°C with presence of a density of asexual stage P. falciparum >100K parasites/µL blood Secondary (10) = >37.5°C with presence of a density of asexual stage P. falciparum >10K parasites/µL blood Secondary (0) = >37.5°C with presence of a density of asexual stage P. falciparum >0 parasites/µL blood Secondary (0*) = >37.5°C OR history of fever in the last 24 hrs with presence of a density of asexual stage P. falciparum >0 parasites/µL blood
Time Frame: starting 14 days after the 3rd vaccination (day 71), every 28 days and ending on day 240
Measure: Number; unit: events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
events
  SA: Primary | 107 | 121
  SA: Secondary (200) | 25 | 29
  SA: Secondary (100) | 68 | 80
  SA: Secondary (10) | 130 | 143
  SA: Secondary (0) | 158 | 165
  SA: Secondary (0*) | 185 | 182
  MT: Primary | 105 | 116
  MT: Secondary (200) | 23 | 27
  MT: Secondary (100) | 64 | 76
  MT: Secondary (10) | 130 | 138
  MT: Secondary (0) | 156 | 161
  MT: Secondary (0*) | 186 | 182
  SA MT: Primary | 101 | 113
  SA MT: Secondary (200) | 22 | 27
  SA MT: Secondary (100) | 60 | 76
  SA MT: Secondary (10) | 125 | 138
  SA MT: Secondary (0) | 151 | 160
  SA MT: Secondary (0*) | 183 | 182

2. Secondary Outcome: Time to First Clinical Episode of P Falciparum Malaria During the Efficacy Follow-up Period Adjusted for Time at Risk - According to Protocol (ATP) Population
Description: Days to first clinical episode of P falciparum malaria during the efficacy f/u period for ATP population
  Time at Risk adjusted for:
  SA= study absence MT= malaria treatment SA MT= study absence and malaria treatment
  Case Definitions:
  Primary = >37.5°C with presence of a density of asexual stage P. falciparum >50K parasites/µL blood Secondary (200) = >37.5°C with presence of a density of asexual stage P. falciparum >200K parasites/µL blood Secondary (100) = >37.5°C with presence of a density of asexual stage P. falciparum >100K parasites/µL blood Secondary (10) = >37.5°C with presence of a density of asexual stage P. falciparum >10K parasites/µL blood Secondary (0) = >37.5°C with presence of a density of asexual stage P. falciparum >0 parasites/µL blood Secondary (0*) = >37.5°C OR history of fever in the last 24 hrs with presence of a density of asexual stage P. falciparum >0 parasites/µL blood
Time Frame: starting 14 days after the 3rd vaccination (day 71), every 28 days and ending on day 240
Measure: Number; unit: events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
events
  SA: Primary | 85 | 86
  SA: Secondary (200) | 17 | 13
  SA: Secondary (100) | 49 | 50
  SA: Secondary (10) | 103 | 107
  SA: Secondary (0) | 130 | 138
  SA: Secondary (0*) | 171 | 168
  MT: Primary | 80 | 79
  MT: Secondary (200) | 16 | 12
  MT: Secondary (100) | 46 | 47
  MT: Secondary (10) | 100 | 101
  MT: Secondary (0) | 127 | 131
  MT: Secondary (0*) | 173 | 168
  SA MT: Primary | 78 | 76
  SA MT: Secondary (200) | 15 | 12
  SA MT: Secondary (100) | 44 | 47
  SA MT: Secondary (10) | 96 | 100
  SA MT: Secondary (0) | 122 | 131
  SA MT: Secondary (0*) | 168 | 168

3. Secondary Outcome: Vaccine-Related Solicited Symptoms During 7-day Follow-up Period by Immunization - Intent to Treat (ITT) Population
Description: Each subject participated in the study approximately 14 months with 7-day follow-up for solicited adverse events (five visits: vaccination day plus post-vaccination days 1, 2, 3, and 6).
  I1 = Immunization 1 I2 = Immunization 2 I3 = Immunization 3
Time Frame: vaccination day plus post-vaccination days 1, 2, 3, and 6
Measure: Number; unit: participants
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
participants
  I1 - Pain | 140 | 9
  I1 - Swelling | 51 | 1
  I1 - Fever | 61 | 11
  I1 - Drowsiness | 1 | 0
  I1 - Loss of appetite | 27 | 6
  I1 - Irritability/fussiness | 14 | 1
  I2 - Pain | 113 | 6
  I2 - Swelling | 28 | 0
  I2 - Fever | 46 | 3
  I2 - Drowsiness | 1 | 0
  I2 - Loss of appetite | 21 | 4
  I2 - Irritability/fussiness | 7 | 0
  I3 - Pain | 66 | 1
  I3 - Swelling | 16 | 1
  I3 - Fever | 17 | 6
  I3 - Drowsiness | 0 | 0
  I3 - Loss of appetite | 5 | 3
  I3 - Irritability/fussiness | 3 | 0

4. Secondary Outcome: Vaccine-Related Solicited Symptoms During 7-day Follow-up Period by Immunization - According to Protocol (ATP) Population
Description: as for outcome 3
Time Frame: vaccination day plus post-vaccination days 1, 2, 3, and 6
Measure: Count of Participants; unit: Participants
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 195 | 190
Participants
  I1 - Pain | 137 | 8
  I1 - Swelling | 50 | 1
  I1 - Fever | 61 | 10
  I1 - Drowsiness | 1 | 0
  I1 - Loss of appetite | 27 | 6
  I1 - Irritability/fussiness | 13 | 1
  I2 - Pain | 113 | 5
  I2 - Swelling | 28 | 0
  I2 - Fever | 46 | 3
  I2 - Drowsiness | 1 | 0
  I2 - Loss of appetite | 21 | 3
  I2 - Irritability/fussiness | 7 | 0
  I3 - Pain | 66 | 1
  I3 - Swelling | 15 | 1
  I3 - Fever | 17 | 6
  I3 - Drowsiness | 0 | 0
  I3 - Loss of appetite | 5 | 3
  I3 - Irritability/fussiness | 3 | 0

5. Secondary Outcome: Vaccine-Related Unsolicited Adverse Events by Immunization - Intent to Treat (ITT) Population
Description: Each subject participated in the study approximately 14 months with 7-day follow-up for solicited adverse events (five visits: vaccination day plus post-vaccination days 1, 2, 3, and 6) and 30-day follow-up for unsolicited events (vaccination day plus 29 subsequent days).
  I1 = Immunization 1 I2 = Immunization 2 I3 = Immunization 3
Time Frame: vaccination day and 29 subsequent days
Population: withdrawals
Measure: Number; unit: adverse events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
adverse events
  I1 - Body as a whole general | 14 | 7
  I2 - Body as a whole general: number analyzed (Participants) | 197 | 196
  I2 - Body as a whole general | 7 | 3
  I3 - Body as a whole general: number analyzed (Participants) | 196 | 191
  I3 - Body as a whole general | 4 | 0
  I1 - History of fever | 13 | 7
  I2 - History of fever: number analyzed (Participants) | 197 | 196
  I2 - History of fever | 7 | 3
  I3 - History of fever: number analyzed (Participants) | 196 | 191
  I3 - History of fever | 4 | 0
  I1 - Fever | 1 | 0
  I2 - Fever: number analyzed (Participants) | 197 | 196
  I2 - Fever | 0 | 0
  I3 - Fever: number analyzed (Participants) | 196 | 191
  I3 - Fever | 0 | 0
  I1 - Rash maculo-papular | 0 | 0
  I2 - Rash maculo-papular: number analyzed (Participants) | 197 | 196
  I2 - Rash maculo-papular | 0 | 0
  I3 - Rash maculo-papular: number analyzed (Participants) | 196 | 191
  I3 - Rash maculo-papular | 1 | 0
  I1 - Gastroenteritis | 0 | 1
  I2 - Gastroenteritis: number analyzed (Participants) | 197 | 196
  I2 - Gastroenteritis | 0 | 0
  I3 - Gastroenteritis: number analyzed (Participants) | 196 | 191
  I3 - Gastroenteritis | 0 | 0
  I1 - Headache | 0 | 0
  I2 - Headache: number analyzed (Participants) | 197 | 196
  I2 - Headache | 0 | 0
  I3 - Headache: number analyzed (Participants) | 196 | 191
  I3 - Headache | 1 | 0
  I1 - Injection site inflammation | 0 | 0
  I2 - Injection site inflammation: number analyzed (Participants) | 197 | 196
  I2 - Injection site inflammation | 0 | 0
  I3 - Injection site inflammation: number analyzed (Participants) | 196 | 191
  I3 - Injection site inflammation | 0 | 1

6. Secondary Outcome: Vaccine-Related Unsolicited Adverse Events by Immunization - According to Protocol (ATP) Population
Description: as for outcome 5
Time Frame: vaccination day and 29 subsequent days
Measure: Number; unit: adverse events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 195 | 190
adverse events
  I1 - Body as a whole general | 13 | 6
  I2 - Body as a whole general | 7 | 2
  I3 - Body as a whole general | 4 | 0
  I1 - History of Fever | 12 | 6
  I2 - History of Fever | 7 | 2
  I3 - History ofFever | 4 | 0
  I1 - Fever | 1 | 0
  I2 - Fever | 0 | 0
  I3 - Fever | 0 | 0
  I1 - Rash maculo-papular | 0 | 0
  I2 - Rash maculo-papular | 0 | 0
  I3 - Rash maculo-papular | 1 | 0
  I1 - Gastroenteritis | 0 | 1
  I2 - Gastroenteritis | 0 | 0
  I3 - Gastroenteritis | 0 | 0
  I1 - Headache | 0 | 0
  I2 - Headache | 0 | 0
  I3 - Headache | 1 | 0
  I1 - Injection site inflammation | 0 | 0
  I2 - Injection site inflammation | 0 | 0
  I3 - Injection site inflammation | 0 | 1

7. Secondary Outcome: Number of Patients Who Showed Symptoms, Unsolicited Adverse Events, and Serious Adverse Events by Immunization
Description: Each subject participated in the study approximately 14 months with 7-day follow-up for solicited adverse events (five visits: vaccination day plus post-vaccination days 1, 2, 3, and 6) and 30-day follow-up for unsolicited events (vaccination day plus 29 subsequent days). Follow-up of SAEs continued for study duration (364 days)
Time Frame: vaccination day plus post-vaccine days 1, 2, 3, and 6; 30 day follow-up for unsolicited events and follow-up for SAEs to continue for duration of study (364 days)
Measure: Number; unit: Number of Participants
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
Number of Participants
  Any solicited symptom | 195 | 85
  Any unsolicited AE | 197 | 197
  Any serious adverse event | 16 | 8
  Red blood cell | 176 | 167
  Resistance mechanism | 167 | 160
  Body as a whole general | 174 | 115
  Skin and appendages | 132 | 132
  Gastroentestinal | 128 | 116
  Application site | 176 | 15
  Respiratory | 61 | 69
  Vision | 36 | 35
  Psychiatric | 30 | 3
  Liver and biliary | 10 | 12
  Central and peripheral nervous system | 12 | 9
  White cell and reticuloendothelial | 6 | 10
  Urinary | 6 | 4
  Platelet bleeding and clotting | 1 | 4
  Musculoskeletal | 1 | 3
  Hearing and vestibular | 1 | 2
  Endocrine | 0 | 2
  Reproductive | 2 | 0

8. Secondary Outcome: Vaccine-Related Local and Systemic Solicited Adverse Events by Immunization - According to Protocol (ATP)
Description: as for outcome 5
Time Frame: vaccination day plus 29 subsequent days
Measure: Number; unit: adverse events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 195 | 190
adverse events
  I1 - Any symptom | 157 | 22
  I1 - Local | 139 | 9
  I1 - Systemic | 82 | 16
  I2 - Any symptom | 131 | 10
  I2 - Local | 113 | 5
  I2 - Systemic | 62 | 6
  I3 - Any symptom | 76 | 10
  I3 - Local | 66 | 1
  I3 - Systemic | 21 | 9

9. Secondary Outcome: Vaccine-Related Local and Systemic Solicited Adverse Events by Immunization - Intent to Treat (ITT)
Description: as for outcome 5
Time Frame: vaccination day plus 29 subsequent days
Measure: Number; unit: adverse events
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
Number analyzed (Participants) | 200 | 200
adverse events
  I1 - Any symptom | 160 | 24
  I1 - Local | 142 | 10
  I1 - Systemic | 83 | 17
  I2 - Any symptom | 131 | 11
  I2 - Local | 113 | 5
  I2 - Systemic | 62 | 7
  I3 - Any symptom | 76 | 10
  I3 - Local | 66 | 1
  I3 - Systemic | 21 | 9

ADVERSE EVENTS:
Time Frame: 14 months to include follow-up for unsolicited adverse events 30 days post dose-3
Arm/Group | FMP1/AS02A | RabAvert (Rabies Vaccine)
All-Cause Mortality (participants affected / at risk) | 1/200 | 0/200
Serious Adverse Events (participants affected / at risk) | 15/200 | 8/200
Other Adverse Events (participants affected / at risk) | 197/200 | 197/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMP1/AS02A (N=200) | RabAvert (Rabies Vaccine) (N=200)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Cerebral malaria; severe anemia (Infections and infestations) | 1 (1) | 1 (1)
Convulsions (Nervous system disorders) | 1 (1) | 1 (1)
Foreign body in ear (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in nostril (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hyper-responsive airway disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1)
Parasitemia >20% (Investigations) | 9 (9) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMP1/AS02A (N=200) | RabAvert (Rabies Vaccine) (N=200)
Malaria (Blood and lymphatic system disorders) | 172 (172) | 166 (166)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
Severe malaria (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Severe anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobinuria (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemai nemolytic (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 167 (167) | 159 (159)
Infection (Infections and infestations) | 2 (2) | 3 (3)
Moniliasis (Infections and infestations) | 4 (4) | 0 (0)
Herpes simplex (Infections and infestations) | 2 (2) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 2 (2)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Skin and subcutaneous tissue disorders) | 66 (66) | 71 (71)
Eczema (Skin and subcutaneous tissue disorders) | 54 (54) | 46 (46)
Dermatitis fungal (Skin and subcutaneous tissue disorders) | 33 (33) | 27 (27)
Otitis media (Skin and subcutaneous tissue disorders) | 8 (8) | 8 (8)
Folliculitis (Skin and subcutaneous tissue disorders) | 6 (6) | 6 (6)
Otitis externa (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Arthropod infestation (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus genital (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Furunculosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Billous eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 39 (39) | 43 (43)
Loss of appetite (anorexia) (Gastrointestinal disorders) | 39 (39) | 41 (41)
Parasitic infection (Gastrointestinal disorders) | 21 (21) | 20 (20)
Gastroenteritis (Gastrointestinal disorders) | 14 (14) | 21 (21)
Abdominal pain (Gastrointestinal disorders) | 13 (13) | 13 (13)
Vomiting (Gastrointestinal disorders) | 13 (13) | 12 (12)
Stomatitis ulcerative (Gastrointestinal disorders) | 6 (6) | 6 (6)
Glossitis (Gastrointestinal disorders) | 6 (6) | 1 (1)
Diarrhea bloody (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Tooth ache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tooth caries (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal rumbling (Gastrointestinal disorders) | 1 (1) | 0 (0)
History of fever (General disorders) | 70 (70) | 61 (61)
Injury (General disorders) | 24 (24) | 28 (28)
Fever (General disorders) | 33 (33) | 16 (16)
Cellulitis (General disorders) | 3 (3) | 7 (7)
Edema (General disorders) | 3 (3) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0)
Abdomen enlarged (General disorders) | 0 (0) | 2 (2)
Varicella (General disorders) | 1 (1) | 0 (0)
Rigors (General disorders) | 1 (1) | 0 (0)
Malnutrion (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Injury (foreign body) (General disorders) | 1 (1) | 0 (0)
Halitosis (General disorders) | 1 (1) | 0 (0)
Face edema (General disorders) | 0 (0) | 1 (1)
Astnenia (General disorders) | 1 (1) | 0 (0)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 33 (33) | 39 (39)
Coughing (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 30 (30)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 36 (36) | 33 (33)
Blepharitis (Immune system disorders) | 1 (1) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 10 (10) | 12 (12)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 4 (4)
Convulsions (Nervous system disorders) | 4 (4) | 3 (3)
Hypokinesia (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Lymphocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 6 (6) | 4 (4)
Urine abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Irritability/fussiness (Psychiatric disorders) | 0 (0) | 1 (1)
Hellucination (Psychiatric disorders) | 1 (1) | 0 (0)
Drowsiness (Psychiatric disorders) | 1 (1) | 0 (0)
Penis disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Weight decrease (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cerumen (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Sialoadenitis (Endocrine disorders) | 0 (0) | 2 (2)
Injection site inflammation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No